CLINICAL TRIAL: NCT07321184
Title: Effect of Polysaccharide-based Complex Administration on the Gut Microbiome and Cardio-Metabolic Profile in Children With Obesity and Metabolic Syndrome.
Acronym: Polymets
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Elvira Verduci, Full Professor, Medical Doctor, University of Milan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/ST/260; Ethical Committe (Other: Comitato Etico Milano Area 1)
Record Dates: First submitted 2025-11-25; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Childhood Obesity
Keywords: childhood obesity; gut microbiota; metabolic syndrome; mediterranean diet; fiber
MeSH Terms: conditions — Pediatric Obesity; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm Pre-Post Treatment (Experimental): At T0 (enrollment), participants will undergo baseline assessments. From T0 to T1, they will receive a polysaccharide-based complex together with a dietary and lifestyle intervention based on Mediterranean diet principles. From T1 to T2, the polysaccharide-based complex will be discontinued, and participants will continue only with the dietary and lifestyle intervention as a washout phase. Assessments at T0, T1, and T2 will be used to evaluate changes over time.
  Interventions: Device: Polysaccharide-based complex

INTERVENTIONS:
Device: Polysaccharide-based complex — The Polysaccharide-based complex is a medical device composed of mixture of soluble and insoluble fibres (cellulose, hemicellulose, pectin, mucilages). After enrolment at T0, participants were instructed to consume a polysaccharide-based complex for 4 months at a dosage of two sachets daily, to be consumed one before lunch and one before dinner (total 5 g/day).
  Other Names: Neo-Policaptil Gel Retard

SUMMARY:
Childhood obesity is a growing public health concern and is associated with long-term health issues. Changing lifestyle habits, especially improving diet and maintaining these changes over time, can be challenging for children and families. For this reason, new treatment options are being explored, including ways to improve the gut microbiota, which can influence appetite and host metabolic health.

This study will investigate the impact of a medical device made of polysaccharide-based complex together with healthy lifestyle and dietary intervention, on gut microbiota composition and metabolic health in children and adolescents with metabolically unhealthy obesity. The study will last 8 months and will include 3 visits: at the start (T0), after 4 months (T1), and after 8 months (T2). From T0 to T1, participants will receive the polysaccharide-based complex along with Mediterranean-style dietary and behavioral intervention. From T1 to T2, only the dietary-lifestyle program will continue.

At each visit, researchers will collect blood samples, perform nutritional and body composition assessment, and collect stool samples to characterise the gut microbiota. The primary aim is to evaluate the effect on gut microbiota composition of a polysaccharide-based complex administration combined with dietary and lifestyle interventions. Furthermore, the study aims to evaluate the effectiveness of this intervention in improving obesity-related parameters and the overall cardiometabolic profile.

ELIGIBILITY:
Inclusion Criteria:

* age 8 to 14 years;
* obesity defined as BMI z-score ≥+2 standard deviation scores (SDS) based on the WHO growth charts
* gestational age 37-42 weeks;
* birth weight >2500 g and <4000 g;
* established condition of MUO, defined as follows:

  1. for children ≤10 years according to the IDEFICS criteria [waist circumference (WC) ≥90th percentile and ≥1 of the followings triglycerides (TG) ≥90th percentile, HDL cholesterol (HDL) ≤10th percentile, systolic blood pressure (SBP) or diastolic blood pressure (DBP) ≥90th percentile, HOMA-insulin resistance ≥90th percentile or fasting glucose ≥90th percentile];
  2. for children >10 years according to the IDF criteria [WC ≥ 90th percentile and ≥1 of the followings TG ≥ 150 mg/Dl, HDL ≤ 40 mg/dL, SBP ≥ 130 mmHg, DBP ≥ 85 mmHg and fasting blood glucose ≥ 100 mg/dl or known Type 2 Diabetes]

Exclusion Criteria:

* diagnosis of secondary obesity;
* treatment with pre/probiotics in the previous 3 months;
* antibiotic treatment in the previous 3 months;
* presence of chronic or acute intestinal disease in the previous 3 months

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
gut microbiota composition | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Collection of fecal samples, bacterial DNA extraction and analysis of V3-V4 hypervariable regions of the prokaryotic 16S ribosomal RNA (rRNA) gene

SECONDARY OUTCOMES:
Body Weight | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Body weight Description: Body weight measured in kilograms using a calibrated scale. Unit of Measure: kg
Height | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Height Description: Standing height measured using a stadiometer. Unit of Measure: cm
Height z-score | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Height z-score Description: Height-for-age z-score calculated according to reference growth charts.
  Unit of Measure: z-score
Body Mass Index | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Body Mass Index (BMI) Description: weight and height will be combined to report BMI in kg/m^2 Unit of measure: kg/m^2
Body Mass Index z-score | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  BMI z-score Description: BMI-for-age z-score calculated according to reference growth charts. Unit of Measure: z-score
Waist circumference | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Waist circumference Description: : Waist circumference measured in centimeters using a non-elastic measuring tape. Unit of Measure: cm
Waist-to-height ratio | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Waist-to-height ratio Description: : Waist-to-height ratio calculated as waist circumference divided by height. Unit of Measure: unitless ratio
Fat mass (kg) | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Total body fat mass expressed in kilograms, assessed using air plethysmography. Unit of Measure: kg
Fat mass (%) | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Percentage of total body fat relative to body weight, assessed using air plethysmography.
  Unit of Measure: %
Fat free mass (kg) | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Total fat-free mass expressed in kilograms, assessed using air plethysmography. Unit of Measure: kg
Fat free mass (%) | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Percentage of fat-free mass relative to body weight, assessed using air plethysmography.
  Unit of Measure: %
Systolic blood pressure | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Systolic blood pressure measured in millimeters of mercury using a calibrated sphygmomanometer.
  Unit of Measure: mmHg
Diastolic blood pressure | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Diastolic blood pressure measured in millimeters of mercury using a calibrated sphygmomanometer.
  Unit of Measure: mmHg
Fasting glucose | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Fasting plasma glucose concentration measured in venous blood samples. Unit of Measure: mg/dL
Fasting insulin | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Fasting plasma insulin concentration measured in venous blood samples. Unit of Measure: µU/mL
Glycated hemoglobin (HbA1c) | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Glycated hemoglobin (HbA1c) concentration measured in whole blood as an indicator of long-term glycemic control.
  Unit of Measure: mmol/mol
Lipid profile | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Fasting serum lipid concentrations including total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides. Each lipid parameter will be analyzed and reported separately.
  Unit of Measure: mg/dL
Liver enzymes | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Serum liver enzyme concentrations including aspartate aminotransferase (AST) and alanine aminotransferase (ALT). Each enzyme will be analyzed and reported separately.
  Unit of Measure: U/L
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Insulin resistance assessed using the Homeostatic Model Assessment of Insulin Resistance (HOMA-IR), calculated from fasting plasma glucose and fasting plasma insulin concentrations.
  Unit of Measure: index value
Quantitative Insulin Sensitivity Check Index (QUICKI) | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Insulin sensitivity assessed using the Quantitative Insulin Sensitivity Check Index (QUICKI), calculated from fasting plasma glucose and fasting plasma insulin concentrations.
  Unit of Measure: index value
Triglyceride-Glucose (TyG) index | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Insulin resistance assessed using the Triglyceride-Glucose (TyG) index, calculated from fasting triglyceride and fasting plasma glucose concentrations.
  Unit of Measure: index value
Atherogenic Index of Plasma (AIP) | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Atherogenic risk assessed using the Atherogenic Index of Plasma (AIP), calculated as the logarithm of the ratio between triglycerides and HDL cholesterol concentrations.
  Unit of Measure: index value
Energy Intake | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Energy intake Unit: kcal/day
Macronutrient intake (grams/day) | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Daily intake of macronutrients expressed in grams per day, including:
  * carbohydrates,
  * sugars,
  * total dietary fibers,
  * insoluble fibers,
  * soluble fibers,
  * proteins,
  * animal proteins,
  * plant proteins,
  * total lipids,
  * saturated fatty acids,
  * monounsaturated fatty acids,
  * polyunsaturated fatty acids, Each macronutrient will be analyzed and reported separately.
  Unit of Measure: g/day
Macronutrient intake (% of energy) | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Contribution of macronutrients to total energy intake expressed as percentage of energy, including:
  * carbohydrates,
  * sugars,
  * proteins,
  * total lipids,
  * saturated fatty acids,
  * monounsaturated fatty acids,
  * polyunsaturated fatty acids,
  * omega-3 fatty acids,
  * omega-6 fatty acids. Each macronutrient will be analyzed and reported separately. Unit of Measure: % of daily energy intake (%En)
Micronutrients (µg/day) | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Daily intake of vitamin B12 and folic acid expressed in micrograms per day. Unit of Measure: µg/day
Micronutrients (mg/day) | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Daily intake of calcium, iron, zinc, and magnesium expressed in milligrams per day.
  Unit of Measure: mg/day
KIDMED score | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Adherence to the Mediterranean diet assessed using the KIDMED questionnaire (score range 0-12).
  Unit of Measure: score

OTHER OUTCOMES:
Mid-upper arm circumference (MUAC) | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Mid-upper arm circumference (MUAC) Description: : Mid-upper arm circumference measured in centimeters using a non-elastic measuring tape. Unit of Measure: cm
Mid-upper arm circumference (MUAC) z-score | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Mid-upper arm circumference (MUAC) z-score Description: Mid-upper arm circumference-for-age z-score calculated according to reference growth standards. Unit of Measure: z-score
Triceps skinfold thickness | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Triceps skinfold thickness measured in millimeters using a calibrated skinfold caliper.. Unit of Measure: mm
Triceps skinfold thickness z-score | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Triceps skinfold thickness-for-age z-score calculated according to reference growth standards. Unit of Measure: z-score
Presence of MASLD | At enrollment (T0), after 4 months (T1), at the end of the study at 8 months (T2)
  Description: Presence of metabolic dysfunction-associated steatotic liver disease (MASLD) assessed by abdominal ultrasound.
  Measure Type: Dichotomous (Yes/No)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Vittore Buzzi Children's Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared because the study involves minors

REFERENCES:
- [Result] Serra-Majem L, Ribas L, Ngo J, Ortega RM, Garcia A, Perez-Rodrigo C, Aranceta J. Food, youth and the Mediterranean diet in Spain. Development of KIDMED, Mediterranean Diet Quality Index in children and adolescents. Public Health Nutr. 2004 Oct;7(7):931-5. doi: 10.1079/phn2004556. PMID 15482620
- [Result] Altavilla C, Caballero-Perez P. An update of the KIDMED questionnaire, a Mediterranean Diet Quality Index in children and adolescents. Public Health Nutr. 2019 Oct;22(14):2543-2547. doi: 10.1017/S1368980019001058. Epub 2019 May 31. PMID 31146796
- [Result] Stagi S, Lapi E, Seminara S, Pelosi P, Del Greco P, Capirchio L, Strano M, Giglio S, Chiarelli F, de Martino M. Policaptil Gel Retard significantly reduces body mass index and hyperinsulinism and may decrease the risk of type 2 diabetes mellitus (T2DM) in obese children and adolescents with family history of obesity and T2DM. Ital J Pediatr. 2015 Feb 15;41:10. doi: 10.1186/s13052-015-0109-7. PMID 25774705
- [Result] Zimmet P, Alberti KG, Kaufman F, Tajima N, Silink M, Arslanian S, Wong G, Bennett P, Shaw J, Caprio S; IDF Consensus Group. The metabolic syndrome in children and adolescents - an IDF consensus report. Pediatr Diabetes. 2007 Oct;8(5):299-306. doi: 10.1111/j.1399-5448.2007.00271.x. No abstract available. PMID 17850473
- [Result] Ahrens W, Moreno LA, Marild S, Molnar D, Siani A, De Henauw S, Bohmann J, Gunther K, Hadjigeorgiou C, Iacoviello L, Lissner L, Veidebaum T, Pohlabeln H, Pigeot I; IDEFICS consortium. Metabolic syndrome in young children: definitions and results of the IDEFICS study. Int J Obes (Lond). 2014 Sep;38 Suppl 2:S4-14. doi: 10.1038/ijo.2014.130. PMID 25376220
- [Result] Damanhoury S, Newton AS, Rashid M, Hartling L, Byrne JLS, Ball GDC. Defining metabolically healthy obesity in children: a scoping review. Obes Rev. 2018 Nov;19(11):1476-1491. doi: 10.1111/obr.12721. Epub 2018 Aug 28. PMID 30156016